CLINICAL TRIAL: NCT07055620
Title: Effects of Different Dietary Models on Eating Behavior and Obesity Management in Overweight and Obese Individuals: A Randomized Controlled Trial
Brief Title: Effects of Different Dietary Models on Eating Behavior and Obesity Management in Overweight and Obese Individuals
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, SUHİDE BİLGE HORZUM, dietician, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBHORZUM
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Mediterranean Diet; Intermittent Fasting; Diet
Keywords: obesity; Mediterranean diet; intermittent fasting
MeSH Terms: conditions — Intermittent Fasting; Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The numbers assigned to the three different diet groups are as follows. Mediterranean Diet Group
  (1, 2, 6, 9, 13, 15, 18, 22, 24, 26, 29, 33, 37, 39, 41, 44, 47, 49, 52, 58, 63, 66, 69, 71, 75) Standard Diet Group (3, 7, 8, 11, 16, 19, 20, 23, 25, 30, 32, 34, 36, 40, 43, 45, 50, 51, 54, 56, 60, 62, 65, 68, 73 Time-Restricted Eating Group (4, 5, 10, 12, 14, 17, 21, 27, 28, 31, 35, 38, 42, 46, 48, 53, 55, 57, 59, 61, 64, 67, 70, 72, 74)
  Anthropometric measurements of the individuals participating in the study will be taken four times: at the beginning, at the 4th week, at the 8th week and at the 12th week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean diet (Active Comparator): Mediterranean diet
  Interventions: Other: Mediterranean diet
- standard diet and time-restricted feeding (Active Comparator): standard diet and time-restricted feeding
  Interventions: Other: standard diet and time-restricted feeding
- control group (Active Comparator): standard diet
  Interventions: Other: Standard diet

INTERVENTIONS:
Other: Mediterranean diet — The group that will be applied the Mediterranean diet will be prepared with diet lists that include 35-40% carbohydrate, 15-20% protein and 35-45% fat (>50% Monounsaturated Fatty Acid (MUFA)) of daily energy. The Mediterranean diet pyramid will be explained to the participants who will be applied the Mediterranean diet, and the portions and frequency of olive oil, nuts, olives, fish, yogurt, fruits and vegetables that they should consume will be planned by the dietitian. The Mediterranean diet pyramid recommends the frequency of foods that should be consumed daily, weekly and monthly. It recommends consuming fish and seafood at least twice a week, 2 portions of white meat, 2-4 portions of eggs, less than 2 portions of red meat, 1 portion or less of processed meat and less than 3 portions of dessert. It is recommended to consume 2 portions of dairy products, 1-2 portions of oil seeds and nuts, more spices, herbs, garlic and onions on a daily basis.
  Arms: Mediterranean diet
Other: Standard diet — When writing the weight loss diets applied to the individuals in the standard diet group, it will be taken into account that 45-60% of the energy comes from carbohydrates, 10-20% from protein and 20-35% from fat, as specified in the Turkish Nutrition Guide (TUBER). It will be planned that 10% (preferably 7-8%) of the total energy from fat will come from saturated fats (fat found in animal foods, butter, tallow, tail fat), 12-15% from monounsaturated fats (olive oil, hazelnut oil, rapeseed oil) and 7-10% from polyunsaturated fats (corn, soy, sunflower and cottonseed oils containing n-6 fatty acids and fish, fish oil, walnut, flaxseed containing n-3 fatty acids). It will be stated that this ratio is 1 part solid oil, 1 part any vegetable oil and 1.5 or 2 parts olive oil among the oil types.
  Arms: control group
Other: standard diet and time-restricted feeding — In time-restricted nutrition, the focus is on when the food is consumed rather than the type of food. However, in medical nutrition treatment of obesity, the content of the meals is also important along with the time (Soran and Öney 2022). As stated in the Turkish Nutrition Guide (TÜBER), it will be taken into account that 45-60% of the energy comes from carbohydrates, 10-20% from protein and 20-35% from fat (Ministry of Health, 2022). A time-restricted nutrition model will be implemented from intermittent fasting diet models. The time restriction will be planned as 8 hours of eating and 16 hours of fasting, suitable for the lifestyle of the individuals. The feeding time for individuals who agree to participate in the study will be determined as 11.00-12.00 and 19.00-20.00. Individuals will be given 2 main meals and the first meal will start with breakfast or lunch according to their wishes.
  Arms: standard diet and time-restricted feeding

SUMMARY:
The aim of this study is to examine the effects of different diet models (Mediterranean diet, time-restricted feeding and standard diet application) applied to overweight and obese individuals on eating behavior and obesity management.

Sub-objectives can be listed as; Effects of different diet models on body composition, Effects of different diet models on dietary intake, Effects of different diet models on biochemical parameters (such as blood sugar, insulin resistance, lipid profile).

As a result, this study aims to contribute to the development of individualized nutrition counseling programs by determining effective diet strategies in obesity.

DETAILED DESCRIPTION:
Overweight and obesity are among the most significant risk factors for health globally, with more than 1 billion people expected to be obese by 2030. Turkey is projected to be among the countries at high risk of obesity by 2030. Furthermore, obesity is among the preventable risk factors for cardiovascular disease (CVD), cancer, diabetes, stroke, and chronic lung disease, among other noncommunicable diseases (NCDs). Overweight and obesity are widespread and increasing health problems worldwide. Excessive adiposity is associated with insulin resistance, lipid deterioration, and systemic inflammation. A 5-10% weight loss is known to improve metabolic outcomes such as blood sugar, lipid profile, and blood pressure. Individuals employ a variety of strategies to lose weight. Lifestyle interventions that encourage calorie restriction and increased physical activity are the most commonly prescribed interventions by healthcare and clinical practitioners. While continuous energy restriction is a more traditional method for reducing energy intake, intermittent fasting has emerged as a potential alternative in the last decade. Fasting is known as one of the world's oldest traditions and is practiced across various communities for cultural or religious reasons. Fasting has also been used as a treatment for illness in the past. Hippocrates, considered the father of modern medicine, emphasized the importance of fasting during illness with the saying, "Eating when you are sick is feeding your illness." Intermittent fasting (IF), or periods of voluntary abstinence from food and drink, is an ancient practice followed in various forms by many populations worldwide. Intermittent fasting involves fasting or restricting food intake for specific hours of the day or on specific days of the week. IF can be implemented in three different ways: alternate-day fasting, the 5:2 diet, and time-restricted feeding (TRF). Alternate-day fasting involves alternating days of food and drink consumption with days of fasting during which no energy-containing food or drink is consumed. In alternate-day fasting, approximately 20-25% of energy needs are met on fasting days. Modified fasting is also known as the 5:2 method. This eating pattern involves a very low-calorie diet for two non-consecutive days per week, followed by normal energy requirements without energy restriction for the other five days. Another approach, time-restricted feeding (TRF), is used to describe an eating pattern in which food intake is restricted to a time window of 8 hours or less each day. Among intermittent fasting diets, the TRF diet is a lifestyle intervention that restricts food intake to a fixed number of hours. Welton and colleagues reported that the ideal fasting period for positive weight change is 16 hours. In recent years, small-scale human studies demonstrating the importance of time-restricted eating have become widespread. Many of these studies, as in animal studies, have demonstrated the beneficial effects of intermittent fasting on human metabolism. TRF has been found to reduce energy intake, body weight, body fat, blood glucose, triglycerides, glucose tolerance, and inflammatory markers. It has been established that IF may be beneficial in reducing body weight, improving insulin resistance, and reducing infection by regulating circadian rhythms, gut microbial composition, and metabolism. Time-restricted eating has been suggested as a potential weight-loss strategy because it may be more acceptable due to the reduced burden of dietary restriction. Intermittent fasting reduces body fat storage and increases fat mobilization, oxidation, and ketone body production, resulting in weight loss. A study comparing intermittent fasting with low-energy diets found that, although body weight reductions were similar after three months of follow-up, the reduction in fat mass was greater in the intermittent fasting group.

The term "Mediterranean diet" reflects the food combinations typical of Mediterranean populations such as Greeks, Southern Italians, and Spaniards in the early 1960s. Lower rates of cardiovascular disease (CVD) and chronic diseases associated with aging in these populations led to its popularization. Since November 2010, the Mediterranean diet has been included on the list of the Intangible Cultural Heritage of Humanity by UNESCO, as it represents a heritage closely linked to cultures and lifestyles passed down through centuries and is the result of the complex socioeconomic development of Mediterranean populations.

Eating behavior changes from birth onward, depending on many factors. Eating, which is essential for life, can, in some cases, develop into a psychiatric disorder, or differences from normal eating behaviors can occur. Eating is not an automatic process, especially for young people. It is significantly influenced by the cultural, social, and psychological pressures individuals feel. In recent years, various theories have been developed to assess behaviors that can impair eating motivation, adequate food intake, and body weight control. "Emotional eating" refers to eating to cope with negative emotions and relieve stress by ignoring satiety signals without internal physiological hunger signals. "External eating" refers to eating in response to stimuli related to food consumption, regardless of hunger and satiety signals. "Restrictive eating" reflects the degree to which one deliberately restricts food intake.

Today, the prevalence of non-communicable diseases is increasing, and obesity is among the risk factors for these diseases. While many methods are used in the treatment of obesity, the role of medical nutrition therapy is crucial. Various methods are used in medical nutrition therapy for obesity. These methods include the calorie-restricted Mediterranean diet, the time-restricted eating model (a type of intermittent fasting), and standard dietary intervention. This study will evaluate the effects of these dietary models on individuals' body composition, dietary intake, and eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-49 years old
* Having a BMI value between 25 kg/m2- 35 kg/m2
* Not having conditions that impair reality assessment ability and cognitive functions, preventing interviews or filling out scales
* Being literate
* Having a blood test done by a primary care physician within the last seven days
* Agreeing to participate in the study and signing the informed consent form

Exclusion Criteria:

* Pregnant and breastfeeding women,
* Those who could not attend one or more interview sessions,
* Women who have entered menopause,
* Individuals who want to apply another diet model,
* Individuals who have a pacemaker or defibrillator implanted due to the theoretical possibility of interference with device activity due to the current field caused by impedance measurements,
* Those who have any chronic disease and are on a diet,
* Those who regularly use medications that affect metabolism,
* Those who use insulin and oral antidiabetic medications,
* Those who have allergies or intolerances to any food components of the Mediterranean diet (walnuts, hazelnuts, peanuts, almonds, etc.),
* Those who use vitamin/mineral supplements,
* Those who have a psychiatric disease diagnosed by a physician.
* In order to understand the effectiveness of the diet, individuals will be asked to maintain their physical activity levels. Therefore, individuals who want to increase their physical activity levels in addition to the applied diet will not be included in the study.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Diet Satisfaction Scale | 12 weeks
  The validity and reliability study of the scale, originally named "Diet Satisfaction Scale", developed by Jospe and his colleagues in 2020, was conducted by Eskici and his colleagues in 2021 (Jospe et al 2020, Eskici and Yılmaz 2021). The items of the scale, which is used to evaluate issues such as hunger, desire to prepare food, enjoyment of the diet, following the diet at home and away from home, contribution to physical health, food variety, budget suitability and continuity, which affect the satisfaction of the clients with any diet, include 9-item five-point Likert-type (1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree) answer options. Only item 1 is scored in reverse (1=5, 2=4, 3=3, 4=2 and 5=1). The maximum score that can be obtained from the scale is 45. A high score indicates that diet satisfaction increases.
Three Factor Eating Questionnaire (TFEQ-21) | 12 weeks
  In order to determine the eating behavior of the individuals participating in the study, the 21-item Three-Factor Eating Scale, which was validated for Turkish culture by Karakuş et al. in 2016, will be used. All of the items are four-point Likert-type and the answers are as follows; 1= Definitely false, 2= Mostly false, 3= Mostly true and 4= Definitely true. This scale measures eating behavior with three sub-dimensions: cognitive restraint (CRI), uncontrolled eating (URI) and emotional eating (EI). Items 1, 5, 11, 17, 18, and 21 measure CRI and evaluate the tendency to control food intake to maintain body weight and body shape. Items 3, 6, 8, 9, 12, 13, 15, 19, and 20 measure CRI and evaluate the tendency to lose control over eating when hungry and exposed to an external stimulus. EI; Items 2, 4, 7, 10, 14 and 16 measure and evaluate the relationship between a negative mood such as loneliness, demoralization or anxiety and overeating. It is recommended to use the converted scale scor

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Bayrak, Study Director — Selcuk University
Locations (1):
- Eda Ocak Nutrition and Diet Consultancy, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication.
Supporting Information: Study Protocol, ICF
Time Frame: April 2025-November 2025
Access Criteria: Access criteria will be shared with researchers who meet the following conditions:
  Being employed by a recognized academic institution, university, research hospital, or public research organization; Providing documentation that the study in which the requested data will be used has scientific, ethical, and social benefit purposes; Submitting a research protocol approved by the relevant institution or ethics committee; Committing that the data will be used only for secondary analysis or meta-analysis.